CLINICAL TRIAL: NCT02684058
Title: Phase II Open-label Global Study to Evaluate the Effect of Dabrafenib in Combination With Trametinib in Children and Adolescent Patients With BRAF V600 Mutation Positive Low Grade Glioma (LGG) or Relapsed or Refractory High Grade Glioma (HGG)
Brief Title: Study of Efficacy and Safety of Dabrafenib in Combination With Trametinib in Pediatric Patients With BRAF V600 Mutation Positive LGG or Relapsed or Refractory HGG Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDRB436G2201; 2015-004015-20 (EudraCT Number)
Record Dates: First submitted 2016-02-04; First posted 2016-02-17 (Estimated); Results first posted 2023-05-19 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Diffuse Astrocytoma; Anaplastic Astrocytoma; Astrocytoma; Oligodendroglioma, Childhood; Anaplastic Oligodendroglioma; Glioblastoma; Pilocytic Astrocytoma; Giant Cell Astrocytoma; Pleomorphic Xanthoastrocytoma; Anaplastic Pleomorphic Xanthoastrocytoma; Angiocentric Glioma; Chordoid Glioma of Third Ventricle; Gangliocytoma; Ganglioglioma; Anaplastic Ganglioglioma; Dysplastic Gangliocytoma of Cerebrellum; Desmoplastic Infantile Astrocytoma and Ganglioglioma; Papillary Glioneuronal Tumor; Rosette-forming Glioneurona Tumor; Central Neurocytoma; Extraventricular Neurocytoma; Cerebellar Iponeurocytoma
Keywords: Malignant glioma; BRAF mutant positive; High grade glioma; Low grade glioma; Dabrafenib; Trametinib; Pediatrics; Brain neoplasma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Ganglioneuroma; Ganglioglioma; Neurocytoma; Glioma | interventions — dabrafenib; trametinib; Carboplatin; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LGG cohort: dabrafenib and trametinib (Experimental): Participants in the LGG cohort randomized to receive dabrafenib (orally, twice daily and dosed based on weight and age) in combination with trametinib (orally, once daily in combination with the first daily dose of dabrafenib and was dosed based on weight)
  Interventions: Drug: Dabrafenib; Drug: trametinib
- LGG cohort: carboplatin and vincristine (Active Comparator): Participants in the LGG cohort randomized to receive active comparator chemotherapy (carboplatin and vincristine). Participants received one course of induction (10 weeks of chemotherapy with 2 weeks of rest), followed by 8 cycles of maintenance chemotherapy.
  Interventions: Drug: Carboplatin; Drug: Vincristine
- HGG cohort: dabrafenib and trametinib (Experimental): Participants in the HGG cohort received dabrafenib (orally, twice daily and dosed based on weight and age) and trametinib (orally, once daily in combination with the first daily dose of dabrafenib and dosed based on weight)
  Interventions: Drug: Dabrafenib; Drug: trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib was available as 50 mg and 75 mg hard capsules and as 10 mg dispersible tablets for oral suspension. Dabrafenib was administered orally, twice daily, and was dosed based on age and weight Patients < 12 years old and ≥ 16 kg were to be administered either the dabrafenib capsules or dabrafenib dispersible tablets for oral suspension (dose: 5.25 mg/kg/day) Patients ≥ 12 years old and ≥ 19 kg were to be administered either the dabrafenib capsules or dabrafenib dispersible tablets for oral suspension (dose: 4.5 mg/kg/day) Patients < 12 years old and < 16 kg were to be administered dabrafenib dispersible tablets for oral suspension (dose: 5.25 mg/kg/day) Patients ≥12 years old and <19 kg were to be administered dabrafenib dispersible tablets for oral suspension (dose: 4.5 mg/kg/day)
  Other Names: DRB436
  Arms: HGG cohort: dabrafenib and trametinib; LGG cohort: dabrafenib and trametinib
Drug: trametinib — Trametinib was available as 0.5 mg and 2 mg film-coated tablets and as 5.0 mg powder in bottle for oral solution (0.05 mg/ml after reconstitution with 90 ml water).Trametinib was administered orally, once daily in combination with the first daily dose of dabrafenib and was dosed based on age and weight.
  Patients <6 years old and <26 kg were to be administered the trametinib oral solution (dose: 0.032 mg/kg/day) Patients <6 years old and ≥26 kg were to be administered either the trametinib oral solution or trametinib tablets (dose: 0.032 mg/kg/day) Patients ≥6 years old and ≥10 kg < 33 kg were to be administered the trametinib oral solution (dose: 0.025 mg/kg/day) Patients ≥6 years old and ≥33 kg were to be administered either the trametinib oral solution or the trametinib tablets (dose: 0.025 mg/kg/day)
  Other Names: TMT212
  Arms: HGG cohort: dabrafenib and trametinib; LGG cohort: dabrafenib and trametinib
Drug: Carboplatin — Carboplatin was supplied locally as commercially available and labelled accordingly to comply with legal requirements of each country. Carboplatin was administered as one course of induction (10 weeks of chemotherapy with 2 weeks of rest), followed by 8 cycles of maintenance chemotherapy. Each maintenance cycle was 6 weeks, and consisted of 4 weeks of chemotherapy with 2 weeks of rest.
  Induction: 175 mg/m^2 as weekly intravenous (IV) infusion on weeks 1 to 4, and on weeks 7 to 10, on the same day as vincristine dosing Maintenance: 175 mg/m^2 as weekly IV infusion over 60 minutes on weeks 1 to 4 of each cycle.
  Arms: LGG cohort: carboplatin and vincristine
Drug: Vincristine — Vincristine was supplied locally as commercially available and labelled accordingly to comply with legal requirements of each country. Vincristine was administered as one course of induction (10 weeks of chemotherapy with 2 weeks of rest), followed by 8 cycles of maintenance chemotherapy.
  Induction: 1.5 mg/m^2 as weekly IV bolus infusion (0.05 mg/kg if child is <12 kg) (maximum dose of 2.0 mg) for 10 weeks.
  Maintenance: 1.5 mg/m^2 as weekly IV bolus infusion (0.05 mg/kg if child is <12 kg) (maximum dose of 2.0 mg) on weeks 1 to 3 of each cycle, on the same day as carboplatin dosing.
  Arms: LGG cohort: carboplatin and vincristine

SUMMARY:
The purpose of this study was to investigate the activity of dabrafenib in combination with trametinib in children and adolescent patients with BRAF V600 mutation positive low grade glioma (LGG) or relapsed or refractory high grade glioma (HGG)

DETAILED DESCRIPTION:
This study combines two pediatric glioma cohorts (LGG and HGG cohorts) into a multi-center, open-label, Phase II study:

* The LGG cohort is a multi-center, randomized, open-label part of this Phase II study conducted in children and adolescent patients with BRAF V600 mutation-positive LGG whose tumor was unresectable and who required first systemic treatment. Participants in the LGG cohort were randomized in a 2:1 ratio to either dabrafenib plus trametinib or carboplatin with vincristine.
* The HGG cohort is a multi-center, single-arm, open-label part of this Phase II study conducted in children and adolescent patients with BRAF V600 mutation-positive, refractory or relapsed HGG tumors after having received at least one previous standard therapy.

The duration of treatment for participants on dabrafenib plus trametinib in LGG and for all patients in the HGG cohort was continued until the loss of clinical benefit in the opinion of the Investigator, unacceptable toxicity, start of a new anti-neoplastic therapy, discontinuation at the discretion of the investigator or patient/legal guardian, lost to follow-up, death, study termination by the sponsor, or until disease progression. The duration of treatment for patients in the carboplatin with vincristine arm in LGG cohort was continued for the prescribed number of cycles, as tolerated or until unacceptable toxicity, start of a new anti-neoplastic therapy, discontinuation at the discretion of the investigator or patient/legal guardian, lost to follow-up, death, study is terminated by the sponsor or until disease progression. Participants randomized to the carboplatin with vincristine treatment arm were allowed to cross over to receive dabrafenib in combination with trametinib after centrally confirmed RANO-defined disease progression. Crossover was allowed during the treatment period or the post-treatment period.

After discontinuation of study treatment, all participants (LGG and HGG cohorts) were followed for safety for at least 30 days after the last dose of study treatment. All participants who discontinued study treatment for reasons other than disease progression, death, loss to follow up, or withdrawal of consent moved into the post-treatment efficacy follow-up phase. Finally, all participants were followed for survival once they discontinued study treatment for at least 2 years after the last patient first study treatment (except if consent was withdrawn, death, or the patient was lost to follow-up or discontinued study)

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of BRAF V600 mutant High Grade glioma that had relapsed, progressed or failed to respond to frontline therapy
* Diagnosis of BRAF V600 mutant Low Grade glioma with progressive disease following surgical excision, or non-surgical candidates with necessity to begin first systemic treatment because of a risk of neurological impairment with progression.
* Confirmed measurable disease

Key Exclusion Criteria:

* Previous treatment with dabrafenib, trametinib, other RAF inhibitor, other MEK or ERK inhibitor
* HGG patient: Cancer treatment within the past 3 weeks. LGG patient: Any systemic therapy or radiotherapy prior to enrollment
* LGG patients: history of allergic reaction or contraindications to the use of carboplatin or vincristine
* Stem cell transplant within the past 3 months
* History of heart disease
* Pregnant or lactating females

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (56):
- United States (10):
  - Children's Hospital of Orange County, Orange, California
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Nicklaus Childrens Hospital, Miami, Florida
  - Ann and Robert H Lurie Childrens Hospital of Chicago ., Chicago, Illinois
  - Indiana University School of Medicine ., Indianapolis, Indiana
  - Johns Hopkins University IDS Pharmacy John Hopkins Hospital, Baltimore, Maryland
  - Washington University School of Medicine SC, St Louis, Missouri
  - Cincinnati Childrens Hospital Medical Center Cancer & Blood Disease Inst., Cincinnati, Ohio
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children s Hospital Baylor College of Medicine, Houston, Texas
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Australia (2):
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Brussels, Belgium
- Brazil (2):
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Tampere, Finland
- France (6):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (7):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
- Israel (2):
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Litwinsky
- Italy (5):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Japan (3):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Utrecht, CS, Netherlands
- Novartis Investigative Site, Moscow, Russia
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Zurich, Switzerland
- United Kingdom (3):
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Bouffet E, Hansford JR, Garre ML, Hara J, Plant-Fox A, Aerts I, Locatelli F, van der Lugt J, Papusha L, Sahm F, Tabori U, Cohen KJ, Packer RJ, Witt O, Sandalic L, Bento Pereira da Silva A, Russo M, Hargrave DR. Dabrafenib plus Trametinib in Pediatric Glioma with BRAF V600 Mutations. N Engl J Med. 2023 Sep 21;389(12):1108-1120. doi: 10.1056/NEJMoa2303815. PMID 37733309
- [Derived] Hargrave DR, Terashima K, Hara J, Kordes UR, Upadhyaya SA, Sahm F, Bouffet E, Packer RJ, Witt O, Sandalic L, Kieloch A, Russo M, Cohen KJ; Investigators involved in the high-grade glioma cohort. Phase II Trial of Dabrafenib Plus Trametinib in Relapsed/Refractory BRAF V600-Mutant Pediatric High-Grade Glioma. J Clin Oncol. 2023 Nov 20;41(33):5174-5183. doi: 10.1200/JCO.23.00558. Epub 2023 Aug 29. PMID 37643378
- [Derived] Barbato MI, Nashed J, Bradford D, Ren Y, Khasar S, Miller CP, Zolnik BS, Zhao H, Li Y, Bi Y, Shord SS, Amatya AK, Mishra-Kalyani PS, Scepura B, Al-Matari RA, Pazdur R, Kluetz PG, Donoghue M, Singh H, Drezner N. FDA Approval Summary: Dabrafenib in Combination with Trametinib for BRAFV600E Mutation-Positive Low-Grade Glioma. Clin Cancer Res. 2024 Jan 17;30(2):263-268. doi: 10.1158/1078-0432.CCR-23-1503. PMID 37610803
- [Derived] Shahid S, Kushner BH, Modak S, Basu EM, Rubin EM, Gundem G, Papaemmanuil E, Roberts SS. Association of BRAF V600E mutations with vasoactive intestinal peptide syndrome in MYCN-amplified neuroblastoma. Pediatr Blood Cancer. 2021 Oct;68(10):e29265. doi: 10.1002/pbc.29265. Epub 2021 Jul 31. PMID 34331515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 58 centers across 20 countries
Pre-assignment Details: Pediatric patients for both cohorts were screened for eligibility during the 28 days immediately prior to starting study treatment on Day 1.
  In the LGG cohort, 121 patients were screened of whom 110 patients were randomized in a 2:1 ratio to the dabrafenib and trametinib arm or the carboplatin with vincristine arm. 4 participants randomized to chemotherapy arm were never treated.
  In the HGG cohort, 46 patients were screened of whom 41 patients entered the HGG cohort
Groups:
- LGG Cohort: Carboplatin and Vincristine: Participants in the LGG cohort randomized to receive active comparator chemotherapy (carboplatin and vincristine). Participants received one course of induction (10 weeks of chemotherapy with 2 weeks of rest), followed by 8 cycles of maintenance chemotherapy. Participants were allowed to crossover to dabrafenib and trametinib after centrally confirmed and RANO-defined disease progression.
Period: Treatment Period
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine | HGG Cohort: Dabrafenib and Trametinib
Started | 73 | 37 | 41
Treated | 73 | 33 | 41
Completed | 56 | 14 | 17
Not Completed | 17 | 23 | 24
Not completed — Progressive disease | 4 | 10 | 19
Not completed — Adverse Event | 3 | 8 | 1
Not completed — Physician Decision | 5 | 1 | 2
Not completed — New therapy for study indication | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0
Not completed — Subject/guardian decision | 4 | 3 | 0
Not completed — Death | 0 | 0 | 2
Period: Post-treatment Efficacy Follow-up
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine | HGG Cohort: Dabrafenib and Trametinib
Started (Participants who discontinued study treatment for reasons other than disease progression, death, loss to follow up, or withdrawal of consent) | 9 | 22 | 5
Completed | 2 | 14 | 2
Not Completed | 7 | 8 | 3
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Progressive disease | 4 | 3 | 0
Not completed — Subject/guardian decision | 2 | 2 | 0
Not completed — Death | 0 | 0 | 3
Not completed — New therapy for study indication | 0 | 1 | 0
Period: Post-treatment Survival Follow-up
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine | HGG Cohort: Dabrafenib and Trametinib
Started | 11 | 1 | 9
Completed (Alive at the end of the study) | 10 | 1 | 2
Not Completed | 1 | 0 | 7
Not completed — Death | 0 | 0 | 7
Not completed — Lack of Efficacy | 1 | 0 | 0
Period: Crossover Treatment Period
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine | HGG Cohort: Dabrafenib and Trametinib
Started (Participants randomized to the carboplatin with vincristine treatment arm were allowed to cross-over to receive dabrafenib in combination with trametinib treatment after centrally confirmed and RANO-defined disease progression) | 0 | 12 | 0
Completed | 0 | 11 | 0
Not Completed | 0 | 1 | 0
Not completed — Progressive disease | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine | HGG Cohort: Dabrafenib and Trametinib | Total
Number analyzed (Participants) | 73 | 37 | 41 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 73 | 37 | 41 | 151
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 22 | 23 | 89
  Male | 29 | 15 | 18 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 55 | 25 | 25 | 105
  Asian | 5 | 3 | 11 | 19
  Black Or African American | 2 | 3 | 1 | 6
  Not Reported | 2 | 1 | 1 | 4
  Unknown | 6 | 4 | 3 | 13
  Other | 3 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: LGG Cohort: Overall Response Rate (ORR) by Central Independent Assessment Using Response Assessment in Neuro-Oncology (RANO) Criteria
Description: Percentage of participants in the LGG cohort with a best overall confirmed Complete Response (CR) or Partial Response (PR) as assessed per RANO criteria by central independent assessment. The 95% confidence intervals (CIs) were computed using two-sided exact binomial method.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approximately (approx.) 3 years
Population: All participants on the LGG cohort to whom study treatment had been assigned by randomization regardless of whether or not treatment was administered. According to the intent to treat principle, patients were analyzed according to the treatment they had been assigned to during the randomization procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Percentage of participants | 46.6 [34.8 to 58.6] | 10.8 [3.0 to 25.4]
Statistical Analysis 1: Comparison: LGG Cohort: Dabrafenib and Trametinib vs LGG Cohort: Carboplatin and Vincristine; Test type: Superiority — one-sided p-value at 2.5% level of significance; p < 0.001, Chi-squared; Odds Ratio (OR) = 7.19, 95% CI 2-sided [2.3 to 22.4]

2. Primary Outcome: HGG Cohort: Overall Response Rate (ORR) by Central Independent Assessment Using RANO Criteria
Description: Percentage of participants in the HGG cohort with a best overall confirmed CR or PR as assessed per RANO criteria by central independent assessment. The 95% CIs were computed using two-sided exact binomial method.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 3.2 years
Population: All participants on the HGG cohort to whom study treatment had been assigned and who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Percentage of participants | 56.1 [39.7 to 71.5]

3. Secondary Outcome: LGG Cohort: ORR by Investigator Assessment Using RANO Criteria
Description: Percentage of participants in the LGG cohort with a best overall confirmed CR or PR as assessed per RANO criteria by investigator assessment. The 95% CIs were computed using two-sided exact binomial method.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 3 years and up to approx 4.2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Percentage of participants
  Up to approx. 3 years | 54.8 [42.7 to 66.5] | 13.5 [4.5 to 28.8]
  Up to approx. 4.2 years | 58.9 [46.8 to 70.3] | 18.9 [8.0 to 35.2]

4. Secondary Outcome: LGG Cohort: Kaplan-Meier Estimates of Duration of Response (DOR) as Per Central Independent Assessment Using RANO Criteria
Description: Time from first documented response (PR or CR) until disease progression or death as per RANO criteria. Confidence Intervals were estimated using the Brookmeyer Crowley method. Patients who had not progressed or died or had received further anticancer therapy, were censored at the date of the last adequate tumor evaluation.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 3 years and up to approx 4.2 years
Population: Participants on the LGG cohort to whom study treatment had been assigned by randomization regardless of whether or not treatment was administered with a confirmed CR or PR as per central independent review assessment using RANO criteria. According to the intent to treat principle, patients were analyzed according to the treatment they had been assigned to during the randomization procedure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 40 | 6
Months
  Up to approx. 3 years | 20.3 [12.0 to NA] — Not estimable (NA) due to the insufficient number of participants with events | NA [6.6 to NA] — Not estimable (NA) due to the insufficient number of participants with events
  Up to approx 4.2 years | 30.0 [16.6 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 19.4 [6.6 to NA] — Not estimable (NA) due to the insufficient number of participants with events

5. Secondary Outcome: LGG Cohort: Kaplan-Meier Estimates of Duration of Response (DOR) as Per Investigator Assessment Using RANO Criteria
Description: as for outcome 4
Time Frame: Up to approx. 3 years and up to approx 4.2 years
Population: Participants on the LGG cohort to whom study treatment had been assigned by randomization regardless of whether or not treatment was administered with a confirmed CR or PR as per investigator review assessment using RANO criteria. According to the intent to treat principle, patients were analyzed according to the treatment they had been assigned to during the randomization procedure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 43 | 7
Months
  Up to approx. 3 years | NA [25.5 to NA] — Not estimable (NA) due to the insufficient number of participants with events | NA [5.3 to NA] — Not estimable (NA) due to the insufficient number of participants with events
  Up to approx 4.2 years | 44.4 [33.1 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 22.5 [5.3 to NA] — Not estimable (NA) due to the insufficient number of participants with events

6. Secondary Outcome: LGG Cohort: Kaplan-Meier Progression-Free Survival (PFS) as Per Central Independent Assessment Using RANO Criteria
Description: Time from the date of randomization to the date of first documented disease progression as per central independent review assessment using RANO criteria or death due to any cause. Confidence Intervals were estimated using the Brookmeyer Crowley method. Patients who had not progressed or died or had received further anticancer therapy were censored at the date of the last adequate tumor evaluation.
Time Frame: Up to approx. 3 years and up to approx 4.2 years
Population: Participants on the LGG cohort to whom study treatment had been assigned by randomization regardless of whether or not treatment was administered. According to the intent to treat principle, patients were analyzed according to the treatment they had been assigned to during the randomization procedure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Months
  Up to approx. 3 years | 20.1 [12.8 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 7.4 [3.6 to 11.8]
  Up to approx 4.2 years | 24.9 [12.9 to 31.6] | 7.2 [2.8 to 11.2]
Statistical Analysis 1: Comparison: LGG Cohort: Dabrafenib and Trametinib vs LGG Cohort: Carboplatin and Vincristine; Up to approx. 3 years; Test type: Superiority; p < 0.001, Log Rank — Log-rank test at an overall one-sided 2.5% level of significance; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.17 to 0.55]

7. Secondary Outcome: LGG Cohort: Kaplan-Meier Progression-Free Survival (PFS) as Per Investigator Assessment Using RANO Criteria
Description: Time from the date of randomization to the date of first documented disease progression as per investigator assessment using RANO criteria or death due to any cause. Confidence Intervals were estimated using the Brookmeyer Crowley method. Patients who had not progressed or died or had received further anticancer therapy were censored at the date of the last adequate tumor evaluation.
Time Frame: Up to approx. 3 years and up to approx 4.2 years
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Months
  Up to approx. 3 years | NA [NA to NA] — Not estimable (NA) due to the insufficient number of participants with events | NA [12.6 to NA] — Not estimable (NA) due to the insufficient number of participants with events
  Up to approx 4.2 years | 46.0 [38.6 to NA] — Not estimable (NA) due to the insufficient number of participants with events | 30.8 [7.0 to NA] — Not estimable (NA) due to the insufficient number of participants with events

8. Secondary Outcome: LGG Cohort: Kaplan-Meier Estimates of Time to Response (TTR) as Per Central Independent Assessment Using RANO Criteria
Description: Time from randomization to first documented response of CR or PR as per central independent assessment using RANO criteria. CIs were estimated using the Brookmeyer Crowley method. Patients without an event were censored either at the maximum follow-up time (if they experienced disease progression or death), or at their last tumor assessment date.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 4.2 years
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Months | 11.0 [6.0 to NA] — Not estimable (NA) due to the insufficient number of participants with events | NA [NA to NA] — Not estimable (NA) due to the insufficient number of participants with events

9. Secondary Outcome: LGG Cohort: Kaplan-Meier Estimates of Time to Response (TTR) as Per Investigator Assessment Using RANO Criteria
Description: Time from randomization to first documented response of CR or PR as per investigator assessment using RANO criteria. CIs were estimated using the Brookmeyer Crowley method. Patients without an event were censored either at the maximum follow-up time (if they experienced disease progression or death), or at their last tumor assessment date.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 4.2 years
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Months | 7.4 [5.3 to NA] — Not estimable (NA) due to the insufficient number of participants with events | NA [NA to NA] — Not estimable (NA) due to the insufficient number of participants with events

10. Secondary Outcome: LGG Cohort: Clinical Benefit Rate (CBR) by Central Independent Assessment Using RANO Criteria
Description: Percentage of participants with a best overall response of CR or PR, or stable disease (SD) which lasts for 24 weeks or longer.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
  SD: Partient did not qualify for CR, PR, or progressive disease and has stable nonenhancing (T2/FLAIR) lesions on same or lower doses of corticosteroids compared with baseline scan and clinically stable status.
Time Frame: Up to approx. 4.2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Percentage of participants | 86.3 [76.2 to 93.2] | 43.2 [27.1 to 60.5]

11. Secondary Outcome: LGG Cohort: Clinical Benefit Rate (CBR) by Investigator Assessment Using RANO Criteria
Description: as for outcome 10
Time Frame: Up to approx. 4.2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Percentage of participants | 91.8 [83.0 to 96.9] | 56.8 [39.5 to 72.9]

12. Secondary Outcome: LGG Cohort: Kaplan-Meier Estimates of Overall Survival (OS)
Description: Time from first dose to death due to any cause in the LGG cohort. Confidence Intervals were estimated using the Brookmeyer Crowley method. If a patient was not known to have died at the time of analysis cut-off, OS was censored at the date of last contact.
Time Frame: Up to 4.6 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Months | NA [NA to NA] — Not estimable (NA) due to the insufficient number of participants with events | NA [NA to NA] — Not estimable (NA) due to the insufficient number of participants with events

13. Secondary Outcome: LGG Cohort: 2-year OS Estimate
Description: OS was defined as the time from the first dose to death due to any cause in the LGG cohort. The 2-year Kaplan-Meier OS estimate represented the estimated percentage of participants remaining free from OS events for up to 2 years. If a patient was not known to have died at the time of analysis cut-off, OS was censored at the date of last contact
Time Frame: 2 years from first dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Percentage of participants | 100.0 [100.0 to 100.0] | 96.9 [79.8 to 99.6]

14. Secondary Outcome: HGG Cohort: ORR by Investigator Assessment Using RANO Criteria
Description: ORR in the HGG cohort defined as the percentage of participants in the HGG cohort with a best overall confirmed CR or PR as assessed per RANO criteria by investigator assessment. The 95% CIs were computed using two-sided exact binomial method.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 3.2 years and up to approx. 4.8 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Percentage of participants
  Up to approx. 3.2 years | 58.5 [42.1 to 73.7]
  Up to approx. 4.8 years | 61.0 [44.5 to 75.8]

15. Secondary Outcome: HGG Cohort: Kaplan-Meier Estimates of Duration of Response (DOR) as Per Central Independent Assessment Using RANO Criteria
Description: Time from first documented response (PR or CR) until disease progression or death as per central independent assessment using RANO criteria. CIs were estimated using the Brookmeyer Crowley method. Patients who had not progressed or died or had received further anticancer therapy were censored at the date of the last adequate tumor evaluation.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 3.2 years and up to approx. 4.8 years
Population: Participants on the HGG cohort to whom study treatment had been assigned and who received at least one dose of study treatment with a confirmed CR or PR as per central independent assessment using RANO criteria
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 23
Months
  Up to approx. 3.2 years | 22.2 [7.6 to NA] — Not estimable (NA) due to the insufficient number of participants with events
  Up to approx. 4.8 years | 27.4 [9.2 to NA] — Not estimable (NA) due to the insufficient number of participants with events

16. Secondary Outcome: HGG Cohort: Kaplan-Meier Estimates of Duration of Response (DOR) as Per Investigator Assessment Using RANO Criteria
Description: Time from first documented response (PR or CR) until disease progression or death as per investigator assessment using RANO criteria. CIs were estimated using the Brookmeyer Crowley method. Patients who had not progressed or died or had received further anticancer therapy were censored at the date of the last adequate tumor evaluation.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 3.2 years and up to approx. 4.8 years
Population: Participants on the HGG cohort to whom study treatment had been assigned and who received at least one dose of study treatment with a confirmed CR or PR as per investigator assessment using RANO criteria
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 25
Months
  Up to approx. 3.2 years: number analyzed (Participants) | 24
  Up to approx. 3.2 years | 26.6 [14.9 to NA] — Not estimable (NA) due to the insufficient number of participants with events
  Up to approx. 4.8 years | 32.7 [14.9 to NA] — Not estimable (NA) due to the insufficient number of participants with events

17. Secondary Outcome: HGG Cohort: Kaplan-Meier Estimates of Progression Free Survival (PFS) as Per Central Independent Assessment Using RANO Criteria
Description: Time from the date of first dose of study treatment to the date of first documented disease progression as per central independent review assessment using RANO criteria or death due to any cause. Confidence Intervals were estimated using the Brookmeyer Crowley method. Patients who had not progressed or died or had received further anticancer therapy were censored at the date of the last adequate tumor evaluation.
Time Frame: Up to approx. 4.8 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Months | 9.0 [5.3 to 20.1]

18. Secondary Outcome: HGG Cohort: Kaplan-Meier Estimates of Progression Free Survival (PFS) as Per Investigatort Assessment Using RANO Criteria
Description: Time from the date of first dose of study treatment to the date of first documented disease progression as per investigator assessment using RANO criteria or death due to any cause. Confidence Intervals were estimated using the Brookmeyer Crowley method. Patients who had not progressed or died or had received further anticancer therapy were censored at the date of the last adequate tumor evaluation.
Time Frame: Up to approx. 4.8 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Months | 24.0 [12.5 to NA] — Not estimable (NA) due to the insufficient number of participants with events

19. Secondary Outcome: HGG Cohort: Time to Response (TTR) as Per Central Independent Assessment Using RANO Criteria
Description: Time from start of treatment to first documented response of CR or PR as per independent assessment using RANO criteria. CIs were estimated using the Brookmeyer Crowley method. Patients without an event were censored either at the maximum follow-up time (if they experienced disease progression or death), or at their last tumor assessment date.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 4.8 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Months | 8.5 [2.0 to NA] — Not estimable (NA) due to the insufficient number of participants with events

20. Secondary Outcome: HGG Cohort: Time to Response (TTR) as Per Investigator Assessment Using RANO Criteria
Description: Time from start of treatment to first documented response of CR or PR as per investigator assessment using RANO criteria. CIs were estimated using the Brookmeyer Crowley method. Patients without an event were censored either at the maximum follow-up time (if they experienced disease progression or death), or at their last tumor assessment date.
  CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses.
  PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically.
Time Frame: Up to approx. 4.8 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Months | 3.4 [1.8 to NA] — Not estimable (NA) due to the insufficient number of participants with events

21. Secondary Outcome: HGG Cohort: Clinical Benefit Rate (CBR) as Per Central Independent Assessment Using RANO Criteria
Description: as for outcome 10
Time Frame: Up to approx. 4.8 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Percentage of participants | 65.9 [49.4 to 79.9]

22. Secondary Outcome: HGG Cohort: Clinical Benefit Rate (CBR) as Per Investigator Assessment Using RANO Criteria
Description: as for outcome 10
Time Frame: Up to approx. 4.8 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Percentage of participants | 75.6 [59.7 to 87.6]

23. Secondary Outcome: HGG Cohort: Kaplan-Meier Estimates of Overall Survival (OS)
Description: as for outcome 12
Time Frame: Up to 5.1 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Months | NA [19.8 to NA] — Not estimable (NA) due to the insufficient number of participants with events

24. Secondary Outcome: AUClast for Trametinib
Description: Pharmacokinetic (PK) parameters were calculated by standard non-compartmental analysis. AUClast is the area under the curve (AUC) from time zero to the last measurable concentration sampling time (tlast).
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of trametinib with an evaluable AUClast PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (hr) * nanogram (ng)/mililiter (mL)
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 36 | 55
hour (hr) * nanogram (ng)/mililiter (mL) | 282 (53.7) | 328 (33.4)

25. Secondary Outcome: Cmax for Trametinib
Description: PK parameters were calculated by standard non-compartmental analysis. Cmax is the maximum plasma drug concentration after single dose administration
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of trametinib with an evaluable Cmax PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 36 | 55
ng/mL | 21.3 (36.3) | 22.7 (41.1)

26. Secondary Outcome: AUCtau for Trametinib
Description: PK parameters were calculated by standard non-compartmental analysis. AUCtau is the AUC calculated to the end of a dosing interval (tau) at steady-state
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of trametinib with an evaluable AUCtau PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr * ng/mL
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 33 | 44
hr * ng/mL | 307 (22.8) | 339 (22.2)

27. Secondary Outcome: Tmax for Trametinib
Description: PK parameters were calculated by standard non-compartmental analysis. Tmax is the time to reach maximum plasma concentration. Actual recorded sampling times were considered for the calculations.
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of trametinib with an evaluable Tmax PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 36 | 55
hour | 1.67 (58.1) | 1.53 (54.6)

28. Secondary Outcome: T1/2 for Trametinib
Description: PK parameters were calculated by standard non-compartmental analysis. T1/2 is the elimination half-life
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of trametinib with an evaluable T1/2 PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 24 | 14
hour | 26.7 (62.6) | 25.7 (37.9)

29. Secondary Outcome: Ctrough for Trametinib
Description: PK parameters were calculated by standard non-compartmental analysis. Ctrough is the pre-dose plasma concentration
Time Frame: Week 3 Day 1 pre-dose
Population: Participants who received at least one dose of trametinib with an evaluable Ctrough PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 36 | 55
ng/ml | 8.73 (72.7) | 9.82 (30.1)

30. Secondary Outcome: AUClast for Dabrafenib and Its Metabolites (Carboxy-dabrafenib, Desmethyl-dabrafenib Amd Hydroxy-dabrafenib)
Description: PK parameters were calculated by standard non-compartmental analysis. AUClast is the area under the curve (AUC) from time zero to the last measurable concentration sampling time (tlast).
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of dabrafenib with an evaluable AUClast PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr * ng/ml
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 34 | 54
hr * ng/ml
  Dabrafenib | 4330 (44.7) | 4870 (60.3)
  Carboxy-dabrafenib | 73400 (31.5) | 64200 (46.9)
  Desmethyl-dabrafenib | 3520 (60.2) | 3870 (68.2)
  Hydroxy-dabrafenib | 2810 (36.5) | 2980 (50.1)

31. Secondary Outcome: Cmax for Dabrafenib and Its Metabolites (Carboxy-dabrafenib, Desmethyl-dabrafenib Amd Hydroxy-dabrafenib)
Description: as for outcome 25
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of dabrafenib with an evaluable Cmax PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 34 | 54
ng/ml
  Dabrafenib | 1520 (65.9) | 1330 (93.5)
  Carboxy-dabrafenib | 9050 (31.4) | 7210 (51.6)
  Desmethyl-dabrafenib | 388 (67.2) | 377 (67.2)
  Hydroxy-dabrafenib | 801 (58.8) | 687 (82.6)

32. Secondary Outcome: AUCtau for Dabrafenib and Its Metabolites (Carboxy-dabrafenib, Desmethyl-dabrafenib Amd Hydroxy-dabrafenib)
Description: as for outcome 26
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of dabrafenib with an evaluable AUCtau PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr * ng/ml
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 34 | 47
hr * ng/ml
  Dabrafenib | 4300 (44.7) | 4910 (54.0)
  Carboxy-dabrafenib: number analyzed (Participants) | 29 | 47
  Carboxy-dabrafenib | 71200 (34.0) | 60700 (45.7)
  Desmethyl-dabrafenib: number analyzed (Participants) | 27 | 44
  Desmethyl-dabrafenib | 3360 (57.7) | 3660 (66.9)
  Hydroxy-dabrafenib: number analyzed (Participants) | 33 | 47
  Hydroxy-dabrafenib | 2840 (35.7) | 2960 (47.4)

33. Secondary Outcome: Tmax for Dabrafenib and Its Metabolites (Carboxy-dabrafenib, Desmethyl-dabrafenib Amd Hydroxy-dabrafenib)
Description: as for outcome 27
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of dabrafenib with an evaluable Tmax PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 34 | 54
hr
  Dabrafenib | 1.47 (54.2) | 1.47 (52.9)
  Carboxy-dabrafenib | 3.37 (35.4) | 3.66 (51.4)
  Desmethyl-dabrafenib | 2.21 (76.7) | 2.29 (82.0)
  Hydroxy-dabrafenib | 1.97 (45.9) | 1.68 (57.8)

34. Secondary Outcome: T1/2 for Dabrafenib and Its Metabolites (Carboxy-dabrafenib, Desmethyl-dabrafenib Amd Hydroxy-dabrafenib)
Description: PK parameters were calculated by standard non-compartmental analysis. T1/2 is the elimination half-life
Time Frame: Week 3 Day 1 pre-dose and 0.5, 1, 2, 3, 4, 6, 8 hours post-dose
Population: Participants who received at least one dose of dabrafenib with an evaluable T1/2 PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 33 | 18
hr
  Dabrafenib | 2.48 (36.6) | 3.09 (36.4)
  Carboxy-dabrafenib: number analyzed (Participants) | 20 | 8
  Carboxy-dabrafenib | 7.12 (32.3) | 6.59 (43.9)
  Desmethyl-dabrafenib: number analyzed (Participants) | 3 | 1
  Desmethyl-dabrafenib | 7.06 (392.5) | 16.1
  Hydroxy-dabrafenib: number analyzed (Participants) | 20 | 10
  Hydroxy-dabrafenib | 2.66 (47.8) | 3.52 (71.7)

35. Secondary Outcome: Ctrough for Dabrafenib and Its Metabolites (Carboxy-dabrafenib, Desmethyl-dabrafenib Amd Hydroxy-dabrafenib)
Description: PK parameters were calculated by standard non-compartmental analysis. Ctrough is the pre-dose plasma concentration
Time Frame: Week 3 Day 1 pre-dose
Population: Participants who received at least one dose of dabrafenib with an evaluable Ctrough PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 34 | 54
ng/ml
  Dabrafenib | 38.0 (162.0) | 46.0 (125.1)
  Carboxy-dabrafenib | 3980 (46.1) | 3190 (54.4)
  Desmethyl-dabrafenib | 275 (116.5) | 310 (70.1)
  Hydroxy-dabrafenib | 41.8 (123.8) | 44.3 (99.7)

36. Secondary Outcome: HGG and LGG Cohort: Palatability of Dabrafenib Oral Suspension Based on the Palatability Questionnaire Item: Taste of the Medication Before Rinsing the Mouth
Description: Participants who received the dabrafenib dispersible tablets for oral suspension completed a questionnaire to evaluate the palatability of the pediatric formulation. After taking the medication, participants provided feedback on how it tasted before rinsing with water, rating their experience as very good, good, neither good nor bad, bad or very bad. The ratings of very good, good, and neither good nor bad were grouped together for reporting purposes.
Time Frame: Week 1 and Week 5
Population: Participants who received at least one dose of dabrafenib as dispersible tablet for oral suspension and completed the palatability questionnaire for dabrafenib at week 1 or 5.
Measure: Count of Participants; unit: Participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 8 | 32
Participants
  Week 1: Very good, good, and neither good nor bad | 5 | 18
  Week 1: Bad | 2 | 4
  Week 1: Very bad | 0 | 0
  Week 1: Unable to answer question | 0 | 5
  Week 1: Missing | 1 | 5
  Week 5: Very good, good, and neither good nor bad | 6 | 20
  Week 5: Bad | 0 | 1
  Week 5: Very bad | 0 | 1
  Week 5: Unable to answer question | 0 | 2
  Week 5: Missing | 2 | 8

37. Secondary Outcome: HGG and LGG Cohort: Palatability of Trametinib Oral Solution Based on the Palatability Questionnaire Item: Taste of the Medication Before Rinsing the Mouth
Description: Participants who received the trametinib oral solution completed a questionnaire to evaluate the palatability of the pediatric formulation. After taking the medication, participants provided feedback on how it tasted before rinsing with water, rating their experience as very good, good, neither good nor bad, bad or very bad. The ratings of very good, good, and neither good nor bad were grouped together for reporting purposes.
Time Frame: Week 1 and Week 5
Population: Participants who received at least one dose of trametinib oral solution and completed the palatability questionnaire for trametinib at week 1 or 5.
Measure: Count of Participants; unit: Participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 8 | 35
Participants
  Week 1: Very good, good, and neither good nor bad | 2 | 15
  Week 1: Bad | 3 | 5
  Week 1: Very bad | 0 | 2
  Week 1: Unable to answer question | 1 | 4
  Week 1: Missing | 2 | 9
  Week 5: Very good, good, and neither good nor bad | 5 | 12
  Week 5: Bad | 0 | 6
  Week 5: Very bad | 0 | 2
  Week 5: Unable to answer question | 0 | 1
  Week 5: Missing | 3 | 14

38. Secondary Outcome: HGG and LGG Cohort: Palatability of Dabrafenib Oral Suspension Based on the Palatability Assessment: After- Taste Once the Medication Was Swallowed
Description: Participants who received the dabrafenib dispersible tablets for oral suspension completed a questionnaire to evaluate the palatability of the pediatric formulation. After taking the medication, participants provided feedback on the after-taste of the medication after the medication was swallowed, rating their experience as very good, good, neither good nor bad, bad or very bad. The ratings of very good, good, and neither good nor bad were grouped together for reporting purposes.
Time Frame: Week 1 and Week 5
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 8 | 32
Participants
  Week 1: Very good, good, and neither good nor bad | 4 | 13
  Week 1: Bad | 1 | 6
  Week 1: Very bad | 0 | 0
  Week 1: Unable to answer question | 0 | 3
  Week 1: Missing | 3 | 10
  Week 5: Very good, good, and neither good nor bad | 5 | 16
  Week 5: Bad | 0 | 2
  Week 5: Very bad | 0 | 0
  Week 5: Unable to answer question | 0 | 3
  Week 5: Missing | 3 | 11

39. Secondary Outcome: HGG and LGG Cohort: Palatability of Trametinib Oral Solution Based on the Palatability Assessment: After- Taste Once the Medication Was Swallowed
Description: Participants who received the trametinib oral solution completed a questionnaire to evaluate the palatability of the pediatric formulation. After taking the medication, participants provided feedback on the after-taste of the medication after the medication was swallowed, rating their experience as very good, good, neither good nor bad, bad or very bad. The ratings of very good, good, and neither good nor bad were grouped together for reporting purposes.
Time Frame: Week 1 and Week 5
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 8 | 35
Participants
  Week 1: Very good, good, and neither good nor bad | 3 | 15
  Week 1: Bad | 3 | 5
  Week 1: Very bad | 0 | 2
  Week 1: Unable to answer question | 0 | 2
  Week 1: Missing | 2 | 11
  Week 5: Very good, good, and neither good nor bad | 5 | 16
  Week 5: Bad | 0 | 3
  Week 5: Very bad | 0 | 1
  Week 5: Unable to answer question | 0 | 2
  Week 5: Missing | 3 | 13

40. Secondary Outcome: HGG and LGG Cohort: Palatability of Dabrafenib Oral Suspension Based on the Palatability Questionnaire Item: Immediate Reaction Once the Medication Was Placed Into the Mouth
Description: Participants who received the dabrafenib dispersible tablets for oral suspension completed a questionnaire to evaluate the palatability of the pediatric formulation. After taking the medication, participants provided feedback on the immediate reaction once the medication was placed into their mouth, rating their experience as very good, good, neither good nor bad, bad or very bad. The ratings of very good, good, and neither good nor bad were grouped together for reporting purposes.
Time Frame: Week 1 and Week 5
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 8 | 32
Participants
  Week 1: Very good, good, and neither good nor bad | 4 | 13
  Week 1: Bad | 1 | 5
  Week 1: Very bad | 0 | 1
  Week 1: Unable to answer question | 0 | 3
  Week 1: Missing | 3 | 10
  Week 5: Very good, good, and neither good nor bad | 5 | 18
  Week 5: Bad | 0 | 1
  Week 5: Very bad | 0 | 0
  Week 5: Unable to answer question | 0 | 2
  Week 5: Missing | 3 | 11

41. Secondary Outcome: HGG and LGG Cohort: Palatability of Trametinib Oral Solution Based on the Palatability Assessment: Immediate Reaction Once the Medication Was Placed Into the Mouth
Description: Participants who received the trametinib oral solution completed a questionnaire to evaluate the palatability of the pediatric formulation. After taking the medication, participants provided feedback on the immediate reaction once the medication was placed into their mouth, rating their experience as very good, good, neither good nor bad, bad or very bad. The ratings of very good, good, and neither good nor bad were grouped together for reporting purposes.
Time Frame: Week 1 and Week 5
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 8 | 35
Participants
  Week 1: Very good, good, and neither good nor bad | 3 | 15
  Week 1: Bad | 3 | 4
  Week 1: Very Bad | 0 | 3
  Week 1: Unable to answer question | 0 | 2
  Week 1: Missing | 2 | 11
  Week 5: Very good, good, and neither good nor bad | 5 | 15
  Week 5: Bad | 0 | 4
  Week 5: Very Bad | 0 | 2
  Week 5: Unable to answer question | 0 | 1
  Week 5: Missing | 3 | 13

42. Secondary Outcome: HGG and LGG Cohort: Palatability of Dabrafenib Oral Suspension Based on the Palatability Questionnaire Item: Remaining After-taste Once Rinsing the Mouth With Water
Description: Participants who received the dabrafenib dispersible tablets for oral suspension completed a questionnaire to evaluate the palatability of the pediatric formulation. After taking the medication, participants provided feedback on the after-taste of the medication after rinsing with water, rating their experience as very good, good, neither good nor bad, bad or very bad. The ratings of very good, good, and neither good nor bad were grouped together for reporting purposes.
Time Frame: Week 1 and Week 5
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 8 | 32
Participants
  Week 1: Very good, good, and neither good nor bad | 4 | 15
  Week 1: Bad | 2 | 5
  Week 1: Very bad | 0 | 0
  Week 1: Unable to answer question | 1 | 7
  Week 1: Missing | 1 | 5
  Week 5: Very good, good, and neither good nor bad | 6 | 17
  Week 5: Bad | 0 | 2
  Week 5: Very bad | 0 | 1
  Week 5: Unable to answer question | 0 | 4
  Week 5: Missing | 2 | 8

43. Secondary Outcome: HGG and LGG Cohort: Palatability of Trametinib Oral Solution Based on the Palatability Assessment: Remaining After-taste Once Rinsing the Mouth With Water
Description: Participants who received the trametinib oral solution completed a questionnaire to evaluate the palatability of the pediatric formulation. After taking the medication, participants provided feedback on the after-taste of the medication after rinsing with water, rating their experience as very good, good, neither good nor bad, bad or very bad. The ratings of very good, good, and neither good nor bad were grouped together for reporting purposes.
Time Frame: Week 1 and Week 5
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 8 | 35
Participants
  Week 1: Very good, good, and neither good nor bad | 2 | 15
  Week 1: Bad | 2 | 3
  Week 1: Very Bad | 0 | 2
  Week 1: Unable to answer question | 2 | 6
  Week 1: Missing | 2 | 9
  Week 5: Very good, good, and neither good nor bad | 4 | 14
  Week 5: Bad | 0 | 2
  Week 5: Very Bad | 0 | 2
  Week 5: Unable to answer question | 1 | 3
  Week 5: Missing | 3 | 14

44. Secondary Outcome: LGG Cohort: PROMIS Parent Proxy Global Health 7+2 Scores- Global Health Score
Description: The PROMIS Parent Proxy Global Health 7+2 was used to evaluate the quality of life of participants. The questionnaire included 7 items measuring the global health of the patient. 4 items used a 5-level Likert scale with 1=poor and 5=excellent; 1 item used a 5-level Likert scale with 1=never and 5=always; and 2 items used a 5-level Likert scale with 1=never and 5=almost always. The total raw global health score, ranging from 7 to 35, was computed by summing item values, with higher scores indicating better overall well-being. Raw scores were then transformed into T-scores, standardized with a mean of 50 and a standard deviation of 10. Higher T-scores reflected better global health status.
  Participants who discontinued treatment for reasons other than disease progression entered the post-treatment efficacy follow-up phase, where the questionnaire was performed every 16 weeks until disease progression, withdrawal of consent by patient or a parental/legal guardian, or lost to follow-up.
Time Frame: Baseline, and Day 1 of Week 5, 8, 16, 24, 32, 49, 48 and 56, and thereafter every 16 weeks until end of treatment (EOT), EOT, and every 16 weeks in the post-treatment efficacy follow-up phase until disease progression (assessed up to 4.6 years)
Population: All participants on the LGG cohort to whom study treatment had been assigned by randomization (regardless of whether or not treatment was administered) and contributed to this analysis. According to the intent to treat principle, patients were analyzed according to the treatment they had been assigned to during the randomization procedure.
  Number analyzed indicated number of participants with available data for this outcome measure at the specified timepoints.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 61 | 23
Score on a Scale
  Baseline | 42.67 (10.068) | 42.89 (10.502)
  Week 5 Day 1: number analyzed (Participants) | 50 | 18
  Week 5 Day 1 | 42.14 (9.439) | 39.06 (10.109)
  Week 8 Day 1: number analyzed (Participants) | 53 | 18
  Week 8 Day 1 | 43.83 (9.461) | 38.36 (7.759)
  Week 16 Day 1: number analyzed (Participants) | 48 | 10
  Week 16 Day 1 | 44.68 (9.159) | 41.11 (10.798)
  Week 24 Day 1: number analyzed (Participants) | 46 | 10
  Week 24 Day 1 | 45.27 (9.168) | 36.57 (6.241)
  Week 32 Day 1: number analyzed (Participants) | 47 | 11
  Week 32 Day 1 | 45.46 (8.887) | 40.96 (7.159)
  Week 40 Day 1: number analyzed (Participants) | 40 | 7
  Week 40 Day 1 | 45.37 (9.687) | 38.84 (4.960)
  Week 48 Day 1: number analyzed (Participants) | 43 | 10
  Week 48 Day 1 | 44.83 (9.421) | 41.56 (6.953)
  Week 56 Day 1: number analyzed (Participants) | 46 | 7
  Week 56 Day 1 | 44.54 (8.876) | 38.66 (8.851)
  Week 72 Day 1: number analyzed (Participants) | 40 | 0
  Week 72 Day 1 | 44.21 (8.967) |
  Week 88 Day 1: number analyzed (Participants) | 38 | 0
  Week 88 Day 1 | 44.91 (8.847) |
  Week 104 Day 1: number analyzed (Participants) | 39 | 0
  Week 104 Day 1 | 45.60 (8.231) |
  Week 120 Day 1: number analyzed (Participants) | 33 | 0
  Week 120 Day 1 | 44.41 (7.317) |
  Week 136 Day 1: number analyzed (Participants) | 24 | 0
  Week 136 Day 1 | 44.45 (8.074) |
  Week 152 Day 1: number analyzed (Participants) | 17 | 0
  Week 152 Day 1 | 47.88 (10.534) |
  Week 168 Day 1: number analyzed (Participants) | 13 | 0
  Week 168 Day 1 | 46.48 (9.888) |
  EOT: number analyzed (Participants) | 50 | 14
  EOT | 44.98 (10.274) | 39.69 (10.536)
  Post Treatment Follow-Up 1: number analyzed (Participants) | 1 | 4
  Post Treatment Follow-Up 1 | 45.40 | 45.53 (6.288)
  Post Treatment Follow-Up 2: number analyzed (Participants) | 1 | 1
  Post Treatment Follow-Up 2 | 27.70 | 39.70
  Post Treatment Follow-Up 3: number analyzed (Participants) | 1 | 1
  Post Treatment Follow-Up 3 | 43.60 | 34.60
  Post Treatment Follow-Up 4: number analyzed (Participants) | 1 | 2
  Post Treatment Follow-Up 4 | 31.20 | 43.60 (8.061)
  Post Treatment Follow-Up 5: number analyzed (Participants) | 1 | 1
  Post Treatment Follow-Up 5 | 29.40 | 37.90
  Post Treatment Follow-Up 6: number analyzed (Participants) | 0 | 2
  Post Treatment Follow-Up 6 |  | 36.45 (7.425)
  Post Treatment Follow-Up 7: number analyzed (Participants) | 0 | 0
  Post Treatment Follow-Up 8: number analyzed (Participants) | 0 | 1
  Post Treatment Follow-Up 8 |  | 37.90

45. Secondary Outcome: LGG Cohort: PROMIS Parent Proxy Global Health 7+2 Scores- Pain Score
Description: The PROMIS Parent Proxy Global Health 7+2 was used to evaluate the quality of life of participants. The questionnaire included 1 item measuring the pain of the participants. Pain item used a 5-level Likert scale with 1= never and 5= almost always, higher scores indicate worsening pain. Raw scores were then converted into T-scores, standardized with a mean of 50 and a standard deviation of 10. Higher T-scores indicated more severe pain experiences.
  Participants who discontinued treatment for reasons other than disease progression entered the post-treatment efficacy follow-up phase, where the PROMIS Parent Proxy Global 7+2 Health questionnaire was performed every 16 weeks until disease progression, withdrawal of consent by patient or a parental/legal guardian, or lost to follow-up.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 61 | 23
Score on a Scale
  Baseline | 52.14 (7.658) | 52.64 (7.054)
  Week 5 Day 1: number analyzed (Participants) | 51 | 18
  Week 5 Day 1 | 50.11 (7.275) | 50.97 (6.263)
  Week 8 Day 1: number analyzed (Participants) | 54 | 18
  Week 8 Day 1 | 49.93 (7.727) | 51.00 (6.037)
  Week 16 Day 1: number analyzed (Participants) | 48 | 10
  Week 16 Day 1 | 49.72 (7.300) | 51.75 (6.330)
  Week 24 Day 1: number analyzed (Participants) | 46 | 10
  Week 24 Day 1 | 50.65 (7.450) | 51.81 (7.937)
  Week 32 Day 1: number analyzed (Participants) | 47 | 11
  Week 32 Day 1 | 48.77 (6.647) | 49.59 (6.387)
  Week 40 Day 1: number analyzed (Participants) | 40 | 7
  Week 40 Day 1 | 49.87 (6.389) | 52.52 (7.402)
  Week 48 Day 1: number analyzed (Participants) | 43 | 10
  Week 48 Day 1 | 49.89 (6.581) | 51.20 (5.903)
  Week 56 Day 1: number analyzed (Participants) | 46 | 7
  Week 56 Day 1 | 48.14 (6.496) | 53.99 (5.466)
  Week 72 Day 1: number analyzed (Participants) | 40 | 0
  Week 72 Day 1 | 49.46 (6.498) |
  Week 88 Day 1: number analyzed (Participants) | 38 | 0
  Week 88 Day 1 | 47.82 (6.083) |
  Week 104 Day 1: number analyzed (Participants) | 39 | 0
  Week 104 Day 1 | 48.74 (6.605) |
  Week 120 Day 1: number analyzed (Participants) | 33 | 0
  Week 120 Day 1 | 48.56 (7.583) |
  Week 136 Day 1: number analyzed (Participants) | 24 | 0
  Week 136 Day 1 | 46.16 (5.305) |
  Week 152 Day 1: number analyzed (Participants) | 17 | 0
  Week 152 Day 1 | 47.42 (6.765) |
  Week 168 Day 1: number analyzed (Participants) | 13 | 0
  Week 168 Day 1 | 48.61 (6.298) |
  EOT: number analyzed (Participants) | 50 | 14
  EOT | 51.46 (6.830) | 52.87 (6.113)
  Post Treatment Follow-Up 1: number analyzed (Participants) | 1 | 4
  Post Treatment Follow-Up 1 | 53.05 | 50.60 (4.900)
  Post Treatment Follow-Up 2: number analyzed (Participants) | 1 | 1
  Post Treatment Follow-Up 2 | 58.51 | 43.25
  Post Treatment Follow-Up 3: number analyzed (Participants) | 1 | 1
  Post Treatment Follow-Up 3 | 53.05 | 43.25
  Post Treatment Follow-Up 4: number analyzed (Participants) | 1 | 2
  Post Treatment Follow-Up 4 | 58.51 | 43.25 (0.000)
  Post Treatment Follow-Up 5: number analyzed (Participants) | 1 | 1
  Post Treatment Follow-Up 5 | 58.51 | 43.25
  Post Treatment Follow-Up 6: number analyzed (Participants) | 0 | 2
  Post Treatment Follow-Up 6 |  | 50.88 (10.790)
  Post Treatment Follow-Up 7: number analyzed (Participants) | 0 | 0
  Post Treatment Follow-Up 8: number analyzed (Participants) | 0 | 1
  Post Treatment Follow-Up 8 |  | 43.25

46. Secondary Outcome: LGG Cohort: PROMIS Parent Proxy Global Health 7+2 Scores- Fatigue Score
Description: The PROMIS Parent Proxy Global Health 7+2 was used to evaluate the quality of life of participants. The questionnaire included 1 item measuring the fatigue interference of the participants. Fatigue item used a 5-level Likert scale with 1= never and 5= almost always, higher scores indicate worsening fatigue. Raw scores were then converted into T-scores, standardized with a mean of 50 and a standard deviation of 10. Higher T-scores indicated a greater level of reported fatigue.
  Participants who discontinued treatment for reasons other than disease progression entered the post-treatment efficacy follow-up phase, where the PROMIS Parent Proxy Global 7+2 Health questionnaire was performed every 16 weeks until disease progression, withdrawal of consent by patient or a parental/legal guardian, or lost to follow-up.
Time Frame: as for outcome 44
Population: All participants on the LGG cohort to whom study treatment had been assigned by randomization regardless of whether or not treatment was administered and contributed to this analysis. According to the intent to treat principle, patients were analyzed according to the treatment they had been assigned to during the randomization procedure. Number analyzed indicated number of participants with available data for this outcome measure at the specified timepoints.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 61 | 23
Score on a Scale
  Baseline | 53.30 (6.731) | 54.37 (7.981)
  Week 5 Day 1: number analyzed (Participants) | 51 | 18
  Week 5 Day 1 | 53.96 (7.588) | 56.88 (6.430)
  Week 8 Day 1: number analyzed (Participants) | 54 | 18
  Week 8 Day 1 | 52.68 (6.967) | 58.10 (4.823)
  Week 16 Day 1: number analyzed (Participants) | 48 | 10
  Week 16 Day 1 | 51.22 (6.983) | 57.81 (6.193)
  Week 24 Day 1: number analyzed (Participants) | 46 | 10
  Week 24 Day 1 | 51.04 (8.005) | 55.02 (7.248)
  Week 32 Day 1: number analyzed (Participants) | 47 | 11
  Week 32 Day 1 | 52.49 (7.219) | 57.66 (5.899)
  Week 40 Day 1: number analyzed (Participants) | 40 | 7
  Week 40 Day 1 | 52.27 (7.450) | 58.49 (7.072)
  Week 48 Day 1: number analyzed (Participants) | 43 | 10
  Week 48 Day 1 | 51.65 (7.362) | 53.48 (8.004)
  Week 56 Day 1: number analyzed (Participants) | 46 | 7
  Week 56 Day 1 | 50.51 (7.150) | 57.63 (7.254)
  Week 72 Day 1: number analyzed (Participants) | 40 | 0
  Week 72 Day 1 | 49.93 (6.910) |
  Week 88 Day 1: number analyzed (Participants) | 38 | 0
  Week 88 Day 1 | 50.52 (7.358) |
  Week 104 Day 1: number analyzed (Participants) | 39 | 0
  Week 104 Day 1 | 51.11 (6.899) |
  Week 120 Day 1: number analyzed (Participants) | 33 | 0
  Week 120 Day 1 | 50.40 (7.317) |
  Week 136 Day 1: number analyzed (Participants) | 24 | 0
  Week 136 Day 1 | 50.97 (8.667) |
  Week 152 Day 1: number analyzed (Participants) | 17 | 0
  Week 152 Day 1 | 47.71 (8.037) |
  Week 168 Day 1: number analyzed (Participants) | 13 | 0
  Week 168 Day 1 | 48.21 (8.188) |
  EOT: number analyzed (Participants) | 50 | 14
  EOT | 52.35 (7.565) | 56.88 (5.246)
  Post Treatment Follow-Up 1: number analyzed (Participants) | 1 | 4
  Post Treatment Follow-Up 1 | 48.94 | 52.36 (6.840)
  Post Treatment Follow-Up 2: number analyzed (Participants) | 1 | 1
  Post Treatment Follow-Up 2 | 62.62 | 62.62
  Post Treatment Follow-Up 3: number analyzed (Participants) | 1 | 1
  Post Treatment Follow-Up 3 | 48.94 | 48.94
  Post Treatment Follow-Up 4: number analyzed (Participants) | 1 | 2
  Post Treatment Follow-Up 4 | 56.07 | 48.94 (0.000)
  Post Treatment Follow-Up 5: number analyzed (Participants) | 1 | 1
  Post Treatment Follow-Up 5 | 62.62 | 48.94
  Post Treatment Follow-Up 6: number analyzed (Participants) | 0 | 2
  Post Treatment Follow-Up 6 |  | 55.78 (9.673)
  Post Treatment Follow-Up 7: number analyzed (Participants) | 0 | 0
  Post Treatment Follow-Up 8: number analyzed (Participants) | 0 | 1
  Post Treatment Follow-Up 8 |  | 48.94

47. Post Hoc Outcome: All-collected Deaths
Description: On-treatment deaths were collected from 1st dose to 30 days after last dose of treatment (or start of crossover treatment), up to 4.2 years (LGG) and 4.1 years (HGG). Post- treatment (efficacy/survival) follow-up deaths were collected from 31 days post-treatment to end of study (or start of crossover treatment), up to 4.6 years (LGG) and 5.1 years (HGG). For participants in the LGG cohort who crossed over to dabrafenib and trametinib, on-treatment deaths were collected from 1st dose to 30 days after last dose of crossover treatment, up to 4.2 years. None of the patients who crossed-over were included in the crossover post-treatment efficacy/survival follow-up.
Time Frame: On-treatment: Up to 4.2 years (LGG) and 4.1 years (HGG). Post- treatment: Up to 4.6 years (LGG) and 5.1 years (HGG).Crossover arm: on-treatment: up to 4.2 years
Population: Safety set including all participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 73 | 33 | 41
Participants
  On- treatment deaths | 0 | 0 | 6
  Post-treatment efficacy/survival follow-up deaths: number analyzed (Participants) | 11 | 16 | 13
  Post-treatment efficacy/survival follow-up deaths | 0 | 0 | 11
  Crossover on-treatment deaths: number analyzed (Participants) | 0 | 12 | 0
  Crossover on-treatment deaths |  | 1 |
  Crossover post-treatment efficacy/survival follow-up deaths: number analyzed (Participants) | 0 | 0 | 0
  Crossover post-treatment efficacy/survival follow-up deaths | 0 | 0 | 0
  All deaths | 0 | 1 | 17

48. Other Pre Specified Outcome: LGG Cohort: Overall Response Rate (ORR) by Central Independent Assessment Using RANO Criteria (Longer Follow-up Time)
Description: Percentage of participants with a best overall confirmed CR or PR as assessed per RANO criteria by central independent assessment. The 95% CIs were computed using two-sided exact binomial method. CR: Complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; no new lesions; and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be off steroids or only on physiologic replacement doses. PR: ≥ 50% reduction, compared to baseline, in the sum of products of the perpendicular diameters for all measurable lesions for at least 4 weeks, no progression of nonmeasureable disease, no new lesions, and stable or improved nonenhancing (T2/FLAIR) lesions. Patient must be on a corticosteroid dose not greater than the dose at the time of baseline scan and be stable or improving clinically. This analysis was conducted at the end of the trial (after the primary endpoint analysis cut-off date) and includes a longer follow-up time
Time Frame: Up to approx 4.2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LGG Cohort: Dabrafenib and Trametinib | LGG Cohort: Carboplatin and Vincristine
Number analyzed (Participants) | 73 | 37
Percentage of participants | 54.8 [42.7 to 66.5] | 16.2 [6.2 to 32.0]

49. Other Pre Specified Outcome: HGG Cohort: Overall Response Rate (ORR) by Central Independent Assessment Using RANO Criteria (Longer Follow-up Time)
Description: as for outcome 48
Time Frame: Up to approx 4.8 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HGG Cohort: Dabrafenib and Trametinib
Number analyzed (Participants) | 41
Percentage of participants | 56.1 [39.7 to 71.5]

ADVERSE EVENTS:
Time Frame: On-treatment AEs: from first dose to 30 days after last dose of treatment (or start of crossover treatment), up to 4.2 years (LGG) and 4.1 years (HGG). Post- treatment deaths: from 31 days post-treatment to end of study (or start of crossover treatment), up to 4.6 years (LGG) and 5.1 years (HGG).Crossover on-treatment: AEs from first dose to 30 days after last dose of crossover treatment, up to 4.2 years.
Description: Deaths in the post treatment follow-up period are not considered Adverse Events. The total number at risk in the post treatment includes patients that entered the post treatment follow-up period (post-treatment efficacy and/or survival follow-up). Analysis performed in the safety set including participants who received at least one dose of study treatment. None of the patients who crossed-over were included in the crossover post-treatment efficacy/survival follow-up.
Groups:
- HGG Cohort: Dabrafenib and Trametinib (On-treatment): AEs collected during on-treatment period with dabrafenib and trametinib in the HGG cohort (up to 30 days post- treatment)
- HGG Cohort: Dabrafenib and Trametinib (Post-treatment Follow-up): Deaths collected in the post- treatment follow-up period for participants in the HGG cohort treated with dabrafenib and trametinib (starting from day 31 post- treatment). No AEs were collected during this period
- LGG Cohort: Dabrafenib and Trametinib (On-treatment): AEs collected during on-treatment period with dabrafenib and trametinib in the LGG cohort (up to 30 days post- treatment)
- LGG Cohort: Dabrafenib and Trametinib (Post-treatment Follow-up): Deaths collected in the post- treatment follow-up period for participants in the LGG cohort treated with dabrafenib and trametinib (starting from day 31 post- treatment). No AEs were collected during this period
- LGG Cohort: Carboplatin and Vincristine (On-treatment): AEs collected during on-treatment period with carboplatin and vincristine in the LGG cohort (up to 30 days post- treatment or start date of crossover treatment, whichever was earlier)
- LGG Cohort: Carboplatin and Vincristine (Post-treatment Follow-up): Deaths collected in the post- treatment follow-up period (starting from day 31 post- treatment) for participants in the LGG cohort treated with carboplatin and vincristine. No AEs were collected during this period
- LGG Cohort: Carboplatin and Vincristine (Crossover On-treatment): AEs collected during crossover on-treatment period with dabrafenib and trametinib for participants in the LGG cohort randomized to carboplatin and vincristine who crossedover to dabrafenib and trametinib after disease progression (up to 30 days post- crossover treatment)
- LGG Cohort: Carboplatin and Vincristine (Crossover Post-treatment Follow-up): Deaths collected in the crossover post- treatment follow-up period (starting from day 31 post- crossover treatment) for participants in the LGG cohort treated with carboplatin and vincristine who crossed over to dabrafenib and trametinib. No AEs were collected during this period
Arm/Group | HGG Cohort: Dabrafenib and Trametinib (On-treatment) | HGG Cohort: Dabrafenib and Trametinib (Post-treatment Follow-up) | LGG Cohort: Dabrafenib and Trametinib (On-treatment) | LGG Cohort: Dabrafenib and Trametinib (Post-treatment Follow-up) | LGG Cohort: Carboplatin and Vincristine (On-treatment) | LGG Cohort: Carboplatin and Vincristine (Post-treatment Follow-up) | LGG Cohort: Carboplatin and Vincristine (Crossover On-treatment) | LGG Cohort: Carboplatin and Vincristine (Crossover Post-treatment Follow-up)
All-Cause Mortality (participants affected / at risk) | 6/41 | 11/13 | 0/73 | 0/11 | 0/33 | 0/16 | 1/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 28/41 | 0/0 | 34/73 | 0/0 | 14/33 | 0/0 | 4/12 | 0/0
Other Adverse Events (participants affected / at risk) | 41/41 | 0/0 | 73/73 | 0/0 | 33/33 | 0/0 | 11/12 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | HGG Cohort: Dabrafenib and Trametinib (On-treatment) (N=41) | HGG Cohort: Dabrafenib and Trametinib (Post-treatment Follow-up) (N=0) | LGG Cohort: Dabrafenib and Trametinib (On-treatment) (N=73) | LGG Cohort: Dabrafenib and Trametinib (Post-treatment Follow-up) (N=0) | LGG Cohort: Carboplatin and Vincristine (On-treatment) (N=33) | LGG Cohort: Carboplatin and Vincristine (Post-treatment Follow-up) (N=0) | LGG Cohort: Carboplatin and Vincristine (Crossover On-treatment) (N=12) | LGG Cohort: Carboplatin and Vincristine (Crossover Post-treatment Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Ventricular enlargement (Cardiac disorders) | 0 | NA | 1 | NA | 0 | NA | 0/9 | NA
Detachment of retinal pigment epithelium (Eye disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Ascites (Gastrointestinal disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Constipation (Gastrointestinal disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Pancreatitis (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Vomiting (Gastrointestinal disorders) | 1 | NA | 3 | NA | 0 | NA | 0 | NA
General physical health deterioration (General disorders) | 2 | NA | 0 | NA | 0 | NA | 0/9 | NA
Influenza like illness (General disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Malaise (General disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Pain (General disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Pyrexia (General disorders) | 3 | NA | 12 | NA | 6 | NA | 2 | NA
Bacterial sepsis (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Brain abscess (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Bronchitis (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Device related infection (Infections and infestations) | 0 | NA | 1 | NA | 1 | NA | 0 | NA
Encephalomyelitis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Infection (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Laryngitis (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Sepsis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 0/9 | NA
Tonsillitis (Infections and infestations) | 0 | NA | 3 | NA | 0 | NA | 0 | NA
Tooth abscess (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Toxic shock syndrome (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Upper respiratory tract infection (Infections and infestations) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Urinary tract infection (Infections and infestations) | 0 | NA | 2 | NA | 0 | NA | 1 | NA
Urinary tract infection bacterial (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Varicella (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Viral myositis (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Procedural complication (Injury, poisoning and procedural complications) | 0 | NA | 2 | NA | 0 | NA | 0 | NA
Procedural pain (Injury, poisoning and procedural complications) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Tooth avulsion (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
C-reactive protein increased (Investigations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Neutrophil count decreased (Investigations) | 1 | NA | 0 | NA | 0 | NA | 0/9 | NA
Oxygen saturation decreased (Investigations) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Hypernatraemia (Metabolism and nutrition disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Altered state of consciousness (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Cerebral haemorrhage (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Cerebral ventricle dilatation (Nervous system disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Cerebrospinal fluid circulation disorder (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 1 | NA
Depressed level of consciousness (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Dizziness (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Dysarthria (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Facial paralysis (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Headache (Nervous system disorders) | 3 | NA | 1 | NA | 1 | NA | 1 | NA
Hemiparesis (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Hydrocephalus (Nervous system disorders) | 2 | NA | 2 | NA | 0 | NA | 0 | NA
Intracranial pressure increased (Nervous system disorders) | 2 | NA | 0 | NA | 0 | NA | 0 | NA
Ischaemic cerebral infarction (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Migraine with aura (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Paraesthesia (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Paresis (Nervous system disorders) | 1 | NA | 1 | NA | 0 | NA | 0 | NA
Partial seizures (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Peripheral motor neuropathy (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Seizure (Nervous system disorders) | 2 | NA | 2 | NA | 0 | NA | 0 | NA
Agitation (Psychiatric disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Anxiety (Psychiatric disorders) | 1 | NA | 0 | NA | 1 | NA | 0 | NA
Confusional state (Psychiatric disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Mental status changes (Psychiatric disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Renal colic (Renal and urinary disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 2 | NA | 0 | NA | 0 | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | NA | 1 | NA | 0 | NA | 0 | NA
Rash (Skin and subcutaneous tissue disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Embolism (Vascular disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Hypotension (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Papilloedema (Eye disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Haematological infection (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Pneumonia (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Vulvitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Road traffic accident (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Central nervous system lesion (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Optic perineuritis (Nervous system disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Syncope (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Nephrolithiasis (Renal and urinary disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 4.9999% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | HGG Cohort: Dabrafenib and Trametinib (On-treatment) (N=41) | HGG Cohort: Dabrafenib and Trametinib (Post-treatment Follow-up) (N=0) | LGG Cohort: Dabrafenib and Trametinib (On-treatment) (N=73) | LGG Cohort: Dabrafenib and Trametinib (Post-treatment Follow-up) (N=0) | LGG Cohort: Carboplatin and Vincristine (On-treatment) (N=33) | LGG Cohort: Carboplatin and Vincristine (Post-treatment Follow-up) (N=0) | LGG Cohort: Carboplatin and Vincristine (Crossover On-treatment) (N=12) | LGG Cohort: Carboplatin and Vincristine (Crossover Post-treatment Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | NA | 14 | NA | 20 | NA | 0 | NA
Leukopenia (Blood and lymphatic system disorders) | 3 | NA | 3 | NA | 2 | NA | 0 | NA
Lymphopenia (Blood and lymphatic system disorders) | 3 | NA | 0 | NA | 0 | NA | 0 | NA
Neutropenia (Blood and lymphatic system disorders) | 7 | NA | 10 | NA | 10 | NA | 1 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | NA | 1 | NA | 5 | NA | 0 | NA
Aortic valve incompetence (Cardiac disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Vertigo (Ear and labyrinth disorders) | 1 | NA | 4 | NA | 2 | NA | 0 | NA
Eyelid ptosis (Eye disorders) | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 5 | NA | 15 | NA | 7 | NA | 0 | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 | NA | 13 | NA | 2 | NA | 0 | NA
Angular cheilitis (Gastrointestinal disorders) | 3 | NA | 2 | NA | 0 | NA | 1 | NA
Aphthous ulcer (Gastrointestinal disorders) | 1 | NA | 2 | NA | 0 | NA | 1 | NA
Constipation (Gastrointestinal disorders) | 6 | NA | 10 | NA | 12 | NA | 1 | NA
Dental caries (Gastrointestinal disorders) | 1 | NA | 2 | NA | 0 | NA | 1 | NA
Diarrhoea (Gastrointestinal disorders) | 10 | NA | 27 | NA | 6 | NA | 2 | NA
Nausea (Gastrointestinal disorders) | 11 | NA | 21 | NA | 17 | NA | 3 | NA
Stomatitis (Gastrointestinal disorders) | 3 | NA | 6 | NA | 5 | NA | 1 | NA
Vomiting (Gastrointestinal disorders) | 12 | NA | 25 | NA | 17 | NA | 6 | NA
Asthenia (General disorders) | 2 | NA | 2 | NA | 3 | NA | 1 | NA
Catheter site pain (General disorders) | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Chills (General disorders) | 1 | NA | 4 | NA | 1 | NA | 0 | NA
Facial pain (General disorders) | 0 | NA | 1 | NA | 3 | NA | 0 | NA
Fatigue (General disorders) | 6 | NA | 25 | NA | 10 | NA | 1 | NA
Influenza like illness (General disorders) | 1 | NA | 1 | NA | 2 | NA | 0 | NA
Oedema peripheral (General disorders) | 4 | NA | 2 | NA | 0 | NA | 0 | NA
Pyrexia (General disorders) | 20 | NA | 51 | NA | 2 | NA | 7 | NA
Hypersensitivity (Immune system disorders) | 1 | NA | 1 | NA | 6 | NA | 0 | NA
COVID-19 (Infections and infestations) | 6 | NA | 26 | NA | 0 | NA | 3 | NA
Conjunctivitis (Infections and infestations) | 4 | NA | 6 | NA | 2 | NA | 0 | NA
Gingivitis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 1 | NA
Nasopharyngitis (Infections and infestations) | 2 | NA | 9 | NA | 2 | NA | 1 | NA
Otitis media (Infections and infestations) | 1 | NA | 2 | NA | 2 | NA | 0 | NA
Paronychia (Infections and infestations) | 3 | NA | 17 | NA | 0 | NA | 1 | NA
Rash pustular (Infections and infestations) | 1 | NA | 6 | NA | 0 | NA | 1 | NA
Rhinitis (Infections and infestations) | 4 | NA | 7 | NA | 4 | NA | 2 | NA
Sinusitis (Infections and infestations) | 2 | NA | 4 | NA | 0 | NA | 1 | NA
Upper respiratory tract infection (Infections and infestations) | 10 | NA | 16 | NA | 1 | NA | 1 | NA
Urinary tract infection (Infections and infestations) | 3 | NA | 4 | NA | 2 | NA | 1 | NA
Contusion (Injury, poisoning and procedural complications) | 2 | NA | 3 | NA | 3 | NA | 0 | NA
Head injury (Injury, poisoning and procedural complications) | 3 | NA | 1 | NA | 0 | NA | 0 | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | NA | 0 | NA | 5 | NA | 0 | NA
Procedural pain (Injury, poisoning and procedural complications) | 0 | NA | 2 | NA | 2 | NA | 0 | NA
Alanine aminotransferase increased (Investigations) | 4 | NA | 10 | NA | 9 | NA | 2 | NA
Aspartate aminotransferase increased (Investigations) | 3 | NA | 9 | NA | 5 | NA | 3 | NA
Blood alkaline phosphatase increased (Investigations) | 3 | NA | 7 | NA | 1 | NA | 0 | NA
Blood bicarbonate decreased (Investigations) | 0 | NA | 0 | NA | 3 | NA | 0 | NA
Ejection fraction decreased (Investigations) | 4 | NA | 2 | NA | 0 | NA | 0 | NA
Lymphocyte count decreased (Investigations) | 3 | NA | 5 | NA | 5 | NA | 0 | NA
Neutrophil count decreased (Investigations) | 2 | NA | 11 | NA | 16 | NA | 2 | NA
Platelet count decreased (Investigations) | 1 | NA | 4 | NA | 10 | NA | 0 | NA
SARS-CoV-2 test negative (Investigations) | 2 | NA | 4 | NA | 1 | NA | 2 | NA
Weight decreased (Investigations) | 1 | NA | 2 | NA | 4 | NA | 0 | NA
Weight increased (Investigations) | 6 | NA | 12 | NA | 0 | NA | 0 | NA
White blood cell count decreased (Investigations) | 5 | NA | 9 | NA | 12 | NA | 1 | NA
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 | NA | 4 | NA | 8 | NA | 0 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | NA | 2 | NA | 3 | NA | 0 | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | NA | 2 | NA | 2 | NA | 0 | NA
Hypernatraemia (Metabolism and nutrition disorders) | 3 | NA | 3 | NA | 0 | NA | 0 | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | NA | 2 | NA | 4 | NA | 0 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | NA | 3 | NA | 4 | NA | 0 | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | NA | 1 | NA | 6 | NA | 0 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | NA | 2 | NA | 2 | NA | 0 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | NA | 1 | NA | 3 | NA | 1 | NA
Obesity (Metabolism and nutrition disorders) | 0 | NA | 1 | NA | 1 | NA | 1 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | NA | 9 | NA | 1 | NA | 2 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 3 | NA | 7 | NA | 4 | NA | 0 | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | NA | 1 | NA | 2 | NA | 0 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | NA | 7 | NA | 3 | NA | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | NA | 13 | NA | 4 | NA | 1 | NA
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | NA | 1 | NA | 6 | NA | 0 | NA
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | NA | 4 | NA | 0 | NA | 2 | NA
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | NA | 10 | NA | 0 | NA | 1 | NA
Dizziness (Nervous system disorders) | 4 | NA | 8 | NA | 0 | NA | 1 | NA
Headache (Nervous system disorders) | 17 | NA | 39 | NA | 8 | NA | 7 | NA
Neuralgia (Nervous system disorders) | 0 | NA | 0 | NA | 3 | NA | 0 | NA
Paraesthesia (Nervous system disorders) | 3 | NA | 5 | NA | 3 | NA | 0 | NA
Peripheral motor neuropathy (Nervous system disorders) | 0 | NA | 0 | NA | 5 | NA | 0 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | NA | 0 | NA | 5 | NA | 0 | NA
Seizure (Nervous system disorders) | 5 | NA | 4 | NA | 2 | NA | 1 | NA
Device malfunction (Product Issues) | 1 | NA | 0 | NA | 0 | NA | 1 | NA
Anxiety (Psychiatric disorders) | 2 | NA | 1 | NA | 5 | NA | 0 | NA
Intentional self-injury (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Haematuria (Renal and urinary disorders) | 3 | NA | 3 | NA | 2 | NA | 1 | NA
Proteinuria (Renal and urinary disorders) | 1 | NA | 1 | NA | 2 | NA | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | NA | 11 | NA | 4 | NA | 3 | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 2 | NA | 0 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | NA | 16 | NA | 1 | NA | 2 | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | NA | 3 | NA | 2 | NA | 2 | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | NA | 10 | NA | 7 | NA | 4 | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 3 | NA | 2 | NA | 0 | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 2 | NA | 4 | NA | 2 | NA
Acne (Skin and subcutaneous tissue disorders) | 6 | NA | 10 | NA | 0 | NA | 1 | NA
Alopecia (Skin and subcutaneous tissue disorders) | 1 | NA | 2 | NA | 9 | NA | 1 | NA
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | NA | 4 | NA | 0 | NA | 0 | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | NA | 10 | NA | 0 | NA | 2 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 14 | NA | 20 | NA | 1 | NA | 1 | NA
Eczema (Skin and subcutaneous tissue disorders) | 5 | NA | 13 | NA | 0 | NA | 1 | NA
Erythema (Skin and subcutaneous tissue disorders) | 5 | NA | 12 | NA | 0 | NA | 1 | NA
Erythema nodosum (Skin and subcutaneous tissue disorders) | 3 | NA | 5 | NA | 0 | NA | 0 | NA
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | NA | 2 | NA | 0 | NA | 1 | NA
Ingrowing nail (Skin and subcutaneous tissue disorders) | 3 | NA | 2 | NA | 0 | NA | 1 | NA
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | NA | 0 | NA | 1 | NA
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | NA | 6 | NA | 0 | NA | 0 | NA
Papule (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | NA | 0 | NA | 2 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 4 | NA | 9 | NA | 2 | NA | 1 | NA
Rash (Skin and subcutaneous tissue disorders) | 9 | NA | 14 | NA | 3 | NA | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | NA | 13 | NA | 0 | NA | 1 | NA
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | NA | 0 | NA | 1 | NA
Skin striae (Skin and subcutaneous tissue disorders) | 1 | NA | 5 | NA | 0 | NA | 1 | NA
Urticaria (Skin and subcutaneous tissue disorders) | 5 | NA | 6 | NA | 2 | NA | 0 | NA
Hypertension (Vascular disorders) | 3 | NA | 0 | NA | 1 | NA | 0/9 | NA
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Ear pain (Ear and labyrinth disorders) | 1 | NA | 4 | NA | 1 | NA | 1 | NA
Growth hormone deficiency (Endocrine disorders) | 1 | NA | 0 | NA | 0 | NA | 2 | NA
Thyroid disorder (Endocrine disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Dry eye (Eye disorders) | 2 | NA | 4 | NA | 1 | NA | 0 | NA
Eye pain (Eye disorders) | 1 | NA | 3 | NA | 0 | NA | 1 | NA
Uveitis (Eye disorders) | 1 | NA | 4 | NA | 0 | NA | 0 | NA
Vision blurred (Eye disorders) | 1 | NA | 6 | NA | 1 | NA | 1 | NA
Dyspepsia (Gastrointestinal disorders) | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Food poisoning (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Toothache (Gastrointestinal disorders) | 2 | NA | 0 | NA | 0 | NA | 1 | NA
Cyst (General disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Gait disturbance (General disorders) | 0 | NA | 1 | NA | 1 | NA | 1 | NA
Hyperpyrexia (General disorders) | 0 | NA | 1 | NA | 0 | NA | 1 | NA
Malaise (General disorders) | 1 | NA | 2 | NA | 0 | NA | 1 | NA
Non-cardiac chest pain (General disorders) | 2 | NA | 4 | NA | 2 | NA | 2 | NA
Bronchitis (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 1 | NA
Ear infection (Infections and infestations) | 0 | NA | 4 | NA | 0 | NA | 0 | NA
Folliculitis (Infections and infestations) | 1 | NA | 3 | NA | 2 | NA | 0 | NA
Fungal skin infection (Infections and infestations) | 0 | NA | 4 | NA | 0 | NA | 0 | NA
Gastroenteritis (Infections and infestations) | 2 | NA | 4 | NA | 0 | NA | 1 | NA
Oral candidiasis (Infections and infestations) | 1 | NA | 1 | NA | 0 | NA | 1 | NA
Pharyngitis (Infections and infestations) | 1 | NA | 6 | NA | 0 | NA | 0 | NA
Pulpitis dental (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Respiratory tract infection (Infections and infestations) | 1 | NA | 1 | NA | 0 | NA | 1 | NA
Respiratory tract infection viral (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 1 | NA
Tinea manuum (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Tonsillitis (Infections and infestations) | 2 | NA | 2 | NA | 1 | NA | 1 | NA
Vaginal infection (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 1 | NA
Viral infection (Infections and infestations) | 1 | NA | 4 | NA | 0 | NA | 0 | NA
Arthropod bite (Injury, poisoning and procedural complications) | 3 | NA | 2 | NA | 0 | NA | 0 | NA
Ligament sprain (Injury, poisoning and procedural complications) | 2 | NA | 0 | NA | 0 | NA | 1 | NA
Skin abrasion (Injury, poisoning and procedural complications) | 0 | NA | 6 | NA | 1 | NA | 1 | NA
Tibia fracture (Injury, poisoning and procedural complications) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Blood pressure decreased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
SARS-CoV-2 test positive (Investigations) | 0 | NA | 6 | NA | 1 | NA | 0 | NA
Streptococcus test positive (Investigations) | 0 | NA | 1 | NA | 0 | NA | 1 | NA
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | NA | 1 | NA | 0 | NA | 1 | NA
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Ataxia (Nervous system disorders) | 3 | NA | 1 | NA | 0 | NA | 0 | NA
Neuropathy peripheral (Nervous system disorders) | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Presyncope (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 2 | NA
Insomnia (Psychiatric disorders) | 3 | NA | 2 | NA | 1 | NA | 0 | NA
Mental status changes (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Somatic symptom disorder (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | NA | 1 | NA | 2 | NA | 1 | NA
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | NA | 0 | NA | 1 | NA
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | NA | 2 | NA | 0 | NA | 1 | NA
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | NA | 0 | NA | 1 | NA
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | NA | 2 | NA | 2 | NA | 0 | NA
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | NA | 3 | NA | 1 | NA | 1 | NA
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | NA | 4 | NA | 0 | NA | 0 | NA
Rash papular (Skin and subcutaneous tissue disorders) | 0 | NA | 4 | NA | 0 | NA | 0 | NA
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | NA | 4 | NA | 0 | NA | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT02684058/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT02684058/SAP_003.pdf